CLINICAL TRIAL: NCT01329549
Title: An Open-label, Dose Escalation Phase I Study of the Safety and Tolerability of BIBF 1120 in Combination With Carboplatin and Pegylated Liposomal Doxorubicin (PLD) in Japanese Patients With a First, Second or Third Platinum-sensitive Relapse of Advanced Epithelial Ovarian Cancer, Fallopian Tube or Primary Peritoneal Cancer.
Brief Title: Dose Escalation Study of BIBF 1120 in Combination With Carboplatin and PLD in Relapsed Ovarian Cancer (OC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.117
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — nintedanib; 1-dodecylpyridoxal; Culture Media

ARMS (3):
- BIBF 1120 (low) + Carboplatin + PLD (Experimental): BIBF 1120 (low dose) + carboplatin (AUC5 mg/mL*min) + PLD (30 mg/m2)
  Interventions: Drug: BIBF 1120 (low) + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min
- BIBF 1120 (medium) + Carboplatin + PLD (Experimental): BIBF 1120 (medium dose) + carboplatin (AUC5 mg/mL*min) + PLD (30 mg/m2)
  Interventions: Drug: BIBF 1120 (medium) + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min
- BIBF 1120 (high) + Carboplatin + PLD (Experimental): BIBF 1120 (high dose) + carboplatin (AUC5 mg/mL*min) + PLD (30 mg/m2)
  Interventions: Drug: BIBF 1120 (high) + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min

INTERVENTIONS:
Drug: BIBF 1120 (high) + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min — BIBF 1120 twice daily along with standard therapy of PLD + CBDCA
  Arms: BIBF 1120 (high) + Carboplatin + PLD
Drug: BIBF 1120 (medium) + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min — BIBF 1120 twice daily along with standard therapy of PLD + CBDCA
  Arms: BIBF 1120 (medium) + Carboplatin + PLD
Drug: BIBF 1120 (low) + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min — BIBF 1120 twice daily along with standard therapy of PLD + CBDCA
  Arms: BIBF 1120 (low) + Carboplatin + PLD

SUMMARY:
This phase I, open label dose escalation study will investigate the addition of BIBF 1120 to treatment with the combination of carboplatin and Pegylated Liposomal Doxorubicin (PLD) in patients with advanced, platinum sensitive relapsed ovarian cancer, fallopian tube carcinoma or primary peritoneal cancer. Patients will be treated with BIBF 1120 together with carboplatin and PLD in up to 6-9 repeated 28 days treatment courses until disease progression is observed.

ELIGIBILITY:
Inclusion criteria:

1. Female patients, age 20 years or older, with relapse of histologically (on initial diagnosis) confirmed epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal cancer
2. Up to 3 lines of prior chemo therapy, with treatment free interval of >6 months
3. Platinum based chemotherapy in the immediately preceding line.
4. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
5. Written informed consent that is consistent with Good Clinical Practice (GCP) guidelines

Exclusion criteria:

1. Prior chemotherapy with PLD, and any contraindication for therapy with carboplatin or PLD.
2. More than 2 lines of prior therapies that contained angiogenesis inhibitor.
3. Patients for whom surgery is planned, e.g. interval debulking surgery.
4. History of a cerebral vascular accident, transient ischemic attack or subarachnoid haemorrhage within the past 6 months.
5. Serious infections in particular if requiring systemic antibiotic (antimicrobial, antifungal) or antiviral therapy.
6. Laboratory values indicating an increased risk for adverse events.
7. Significant cardiovascular diseases.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Japan (3):
  - 1199.117.003 Boehringer Ingelheim Investigational Site, Akashi, Hyogo
  - 1199.117.002 Boehringer Ingelheim Investigational Site, Chuo-ku,Tokyo
  - 1199.117.001 Boehringer Ingelheim Investigational Site, Hidaka, Saitama

RESULTS

PARTICIPANT FLOW:
Groups:
- Nintedanib (150 mg) + Carboplatin + PLD: Nintedanib (150 mg) was administered orally on day 2 to Day 28 of each cycle + Carboplatin (AUC 5 mg/mL*min) intravenous infusion, day 1, once every 4 weeks + Pegylated liposomal doxorubicin (30 mg/m2) intravenous infusion, day 1, once every 4 weeks
Period: Overall Study
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Treated set: includes all patients who were dispensed study medication and were documented to have received at least 1 dose of study medication.
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) of Nintedanib
Description: to determine the MTD of nintedanib in combination with carboplatin (AUC 5 mg/mL·min) and PLD (30 mg/m2) reflected by the number of DLTs per dose level. This endpoint has not been statistically analyzed in the study report.
Time Frame: 28 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

2. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax)
Description: Cmax was evaluated for nintedanib (BIBF 1120 BS, BIBF 1202 ZW, BIBF 1202 glucuronide), PLD (doxorubicin), and carboplatin (free platinum, total platinum). This endpoint has not been statistically analyzed in the study report.
  Detailed outcome measure time frame:
  total platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31, 46.917,166.917, 334.917, and 502.917 hours after start of infusion of carboplatin in Cycle 1 and 2
  free platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31 hours after start of infusion of carboplatin in Cycle 1 and 2
  PLD: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.75, 3.25, 4.5, 6.5, 8, 9.5, 25, 27, 30, 34, 47.917, 167.917, 335.917, and 503.917 hours after start of infusion of PLD in Cycle 1 and 2
  nintedanib and its metabolites: pre-dose, 1, 2, 3, 4, 6, 8, 10, 23.917 hours after first administration of nintedanib in Cycle 1 and 2
Time Frame: 0.5h after the start of the infusion up to 56 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to the Time of the Last Quantifiable Drug Concentration (AUC0-tz)
Description: AUC0-tz was evaluated for nintedanib (BIBF 1120 BS, BIBF 1202 ZW, BIBF 1202 glucuronide), PLD (doxorubicin), and carboplatin (free platinum, total platinum). Descriptive statistics were not calculated in the study report.
  Detailed outcome measure time frame:
  total platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31, 46.917,166.917, 334.917, and 502.917 hours after start of infusion of carboplatin in Cycle 1 and 2
  free platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31 hours after start of infusion of carboplatin in Cycle 1 and 2
  PLD: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.75, 3.25, 4.5, 6.5, 8, 9.5, 25, 27, 30, 34, 47.917, 167.917, 335.917, and 503.917 hours after start of infusion of PLD in Cycle 1 and 2
  nintedanib and its metabolites: pre-dose, 1, 2, 3, 4, 6, 8, 10, 23.917 hours after first administration of nintedanib in Cycle 1 and 2
Time Frame: 0.5h after the start of the infusion up to 56 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞ was evaluated for nintedanib (BIBF 1120 BS, BIBF 1202 ZW), PLD (doxorubicin), and carboplatin (free platinum, total platinum). Descriptive statistics were not calculated in the study report.
  Detailed outcome measure time frame
  total platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31, 46.917,166.917, 334.917, and 502.917 hours after start of infusion of carboplatin in Cycle 1 and 2
  free platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31 hours after start of infusion of carboplatin in Cycle 1 and 2
  PLD: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.75, 3.25, 4.5, 6.5, 8, 9.5, 25, 27, 30, 34, 47.917, 167.917, 335.917, and 503.917 hours after start of infusion of PLD in Cycle 1 and 2
  nintedanib and its metabolites: pre-dose, 1, 2, 3, 4, 6, 8, 10, 23.917 hours after first administration of nintedanib in Cycle 1 and 2
Time Frame: 0.5h after the start of the infusion up to 56 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

5. Secondary Outcome: Time From Dosing to the Maximum Plasma Concentration (Tmax)
Description: tmax was evaluated for nintedanib (BIBF 1120 BS, BIBF 1202 ZW, BIBF 1202 glucuronide), PLD (doxorubicin), and carboplatin (free platinum, total platinum). Descriptive statistics were not calculated in the study report.
  Detailed outcome measure time frame:
  total platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31, 46.917,166.917, 334.917, and 502.917 hours after start of infusion of carboplatin in Cycle 1 and 2
  free platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31 hours after start of infusion of carboplatin in Cycle 1 and 2
  PLD: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.75, 3.25, 4.5, 6.5, 8, 9.5, 25, 27, 30, 34, 47.917, 167.917, 335.917, and 503.917 hours after start of infusion of PLD in Cycle 1 and 2
  nintedanib and its metabolites: pre-dose, 1, 2, 3, 4, 6, 8, 10, 23.917 hours after first administration of nintedanib in Cycle 1 and 2
Time Frame: 0.5h after the start of the infusion up to 56 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

6. Secondary Outcome: Terminal Half-life (t1/2)
Description: t1/2 was evaluated for nintedanib (BIBF 1120 BS, BIBF 1202 ZW), PLD (doxorubicin), and carboplatin (free platinum, total platinum). Descriptive statistics were not calculated in the study report.
  Detailed outcome measure time frame:
  total platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31, 46.917,166.917, 334.917, and 502.917 hours after start of infusion of carboplatin in Cycle 1 and 2
  free platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31 hours after start of infusion of carboplatin in Cycle 1 and 2
  PLD: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.75, 3.25, 4.5, 6.5, 8, 9.5, 25, 27, 30, 34, 47.917, 167.917, 335.917, and 503.917 hours after start of infusion of PLD in Cycle 1 and 2
  nintedanib and its metabolites: pre-dose, 1, 2, 3, 4, 6, 8, 10, 23.917 hours after first administration of nintedanib in Cycle 1 and 2
Time Frame: 0.5h after the start of the infusion up to 56 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

7. Secondary Outcome: Total Plasma Clearance (CL)
Description: CL was evaluated for doxorubicin, free platinum, total platinum. Descriptive statistics were not calculated in the study report.
  Detailed outcome measure time frame:
  total platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31, 46.917,166.917, 334.917, and 502.917 hours after start of infusion of carboplatin in Cycle 1 and 2
  free platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31 hours after start of infusion of carboplatin in Cycle 1 and 2
  PLD: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.75, 3.25, 4.5, 6.5, 8, 9.5, 25, 27, 30, 34, 47.917, 167.917, 335.917, and 503.917 hours after start of infusion of PLD in Cycle 1 and 2
Time Frame: 0.5h after the start of the infusion up to 56 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

8. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss)
Description: Vss was evaluated for doxorubicin, free platinum, total platinum. Descriptive statistics were not calculated in the study report.
  total platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31, 46.917,166.917, 334.917, and 502.917 hours after start of infusion of carboplatin in Cycle 1 and 2
  free platinum: pre-dose, 0.5, 1, 1.25, 1.75, 2.25, 3.5, 5.5, 7, 8.5, 22.917, 25, 27, 31 hours after start of infusion of carboplatin in Cycle 1 and 2
  PLD: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.75, 3.25, 4.5, 6.5, 8, 9.5, 25, 27, 30, 34, 47.917, 167.917, 335.917, and 503.917 hours after start of infusion of PLD in Cycle 1 and 2
Time Frame: 0.5h after the start of the infusion up to 56 days
Population: Treated set
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first administration of study treatment up to 33 days after the last administration of the study treatment, up to 360 days.
Arm/Group | Nintedanib (150 mg) + Carboplatin + PLD
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (150 mg) + Carboplatin + PLD (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (150 mg) + Carboplatin + PLD (N=2)
Anaemia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The trial was prematurely terminated because of worldwide disruption of pegylated liposomal doxorubicin (PLD) supplies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.